CLINICAL TRIAL: NCT00277147
Title: Salmonella Typhi Vi O-Acetyl Pectin-rEPA Conjugate Vaccine, Phase 1 Trial in Adults at NIH CC
Brief Title: Salmonella Typhi Vi O-Acetyl Pectin-rEPA Conjugate Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060070; 06-CH-0070
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-09-17

CONDITIONS: Typhoid Fever
Keywords: Typhoid Fever; Immunogenicity; Safety; Vaccine; Conjugate; Healthy Volunteer
MeSH Terms: conditions — Typhoid Fever

INTERVENTIONS:
Drug: BB IND 6989

SUMMARY:
This study will evaluate a new (conjugate) vaccine for typhoid fever, which remains a serious disease especially difficult to treat in developing countries. Salmonella typhi, the bacteria causing typhoid fever, have become resistant to several antibiotics increasing the difficulty of treating the disease. The disease may have serious complications effecting bones, brain, and intestines, with permanent injury or death. Methods to control typhoid fever, such as a sanitary water and food supply, along with effective sewage treatment, are not likely to be available soon in those countries.

NIH scientists developed a vaccine called Vi, made of a polysaccharide (a chain of linked sugars) from the surface of Salmonella typhi, the bacteria that cause typhoid fever. It has been approved by the World Health Organization and is licensed in 94 countries. It is effective in adults but not in young children. Clinical trials have shown that chemically binding the Vi to a protein to form a "conjugate vaccine" has improved and extended its efficacy to children (conjugate vaccines to other bacteria, notably meningitis causing bacteria have been used extensively and successfully). Now NIH scientists have developed another vaccine for typhoid fever - using a polysaccharide from fruit, known as pectin. The pectin has been chemically treated so that it resembles Vi. The treated pectin, O-acetyl pectin, is bound to a protein; exoprotein A, (rEPA). The result is a conjugate, as was formed for Vi. Similarly to the Vi conjugate it induces antibodies against Salmonella typhi in laboratory animals. If the O-acetyl pectin conjugate proves successful, it will be evaluated in children ages 5 to 14 years old and in infants, toward using it with routine vaccines for infants.

Volunteers ages 18 to 45 who do not have an allergy to fruit pectin and who have not been vaccinated against nor had typhoid fever within the last 5 years may be eligible for this study.

Volunteers will undergo several tests at their first visit to the clinic for this study. A blood sample (about 2/3 of an ounce) will be taken to test for HIV, hepatitis B and C, complete blood count, liver functions, blood chemistry and pregnancy in women of childbearing age. The blood sample will also be tested for antibodies to Vi, rEPA (the protein of the conjugate), and pectin. There will also be a urine collection for testing. If the laboratory tests are acceptable, volunteers will be asked to return to the clinic on a...

DETAILED DESCRIPTION:
Typhoid fever remains a common, serious and increasingly difficult to treat disease in developing countries. Control measures, such as safe drinking water, and food, and effective sewage, are not likely to be available soon in many of these countries. In the early 1990's most Salmonella typhi from the Mekong Delta region were resistant to chloramphenicol and ampicillin and treatment required new antibiotics such as ciprofloxacin. Now, resistance of S. typhi has spread to ciprofloxacin.

There are three licensed vaccines for typhoid fever. The whole cell parenteral and the oral attenuated vaccines confer only incomplete immunity of limited duration and cannot be incorporated into the routine vaccination of infants. S. typhi capsular polysaccharide (Vi) is safe, easily standardized and only one injection confers about 70% immunity in individuals greater than 5 years of age for at least 3 years. Its immunogenicity is lesser in 2-4 year-olds and it does not elicit protective antibody levels in children less than 2 years-old. Vi does not elicit a booster response at any age (age-related T-cell independent antibody response).

The immunogenicity of Vi is improved by covalently binding it to a protein to form a conjugate. Vi conjugates were safe and more immunogenic than Vi in adults, in 5-14 year-olds and in children 2-4 year-olds, and showed 90% efficacy in the 2-5 year olds for 47 months.

O-acetyl pectin mimics the antigenic properties of Vi. Although not immunogenic alone, O-acetyl pectin when conjugated induces serum Vi antibodies with booster responses in mice and in guinea pigs albeit at slightly lower levels than Vi conjugates in mice. Double immunodiffusion against mouse anti-Vi revealed antigenic identity between O-acetyl pectin and Vi conjugates.

There are advantages to using pectin as the polysaccharide component of conjugate vaccines for typhoid. Pectin is abundant, has no LPS and requires a simple chemical modification to prepare its di-O-acetyl derivative. Our yields of O-acetyl pectin-rEPA were similar to those of Vi-rEPA. Because it may not be reliable to extrapolate data from animals to humans and especially to infants, we propose clinical evaluation of O-acetyl pectin bound to the recombinant protein A of Pseudomonas aeruginosa (rEPA).

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible, volunteers must be 18 to 45 years old, who

1. are not participating in or plan to participate in another research protocol during the next three months;
2. have not been vaccinated against typhoid fever or had typhoid fever within the last 5 years;
3. are not regularly taking a prescription drug for chronic medical condition;
4. have no history of allergy to fruit or fruit pectin;
5. are not pregnant or intend to become pregnant during the study period of 6 months;
6. Whose HIV, HBsAg and HCV tests must be found negative and laboratory tests of liver function, blood chemistry, complete blood count and urine must show no clinically significant abnormality or pregnancy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25
Dates: Start 2006-01-09; Study Completion 2008-09-17

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Szu SC, Bystricky S, Hinojosa-Ahumada M, Egan W, Robbins JB. Synthesis and some immunologic properties of an O-acetyl pectin [poly(1-->4)-alpha-D-GalpA]-protein conjugate as a vaccine for typhoid fever. Infect Immun. 1994 Dec;62(12):5545-9. doi: 10.1128/iai.62.12.5545-5549.1994. PMID 7960137
- [Background] Kossaczka Z, Bystricky S, Bryla DA, Shiloach J, Robbins JB, Szu SC. Synthesis and immunological properties of Vi and di-O-acetyl pectin protein conjugates with adipic acid dihydrazide as the linker. Infect Immun. 1997 Jun;65(6):2088-93. doi: 10.1128/iai.65.6.2088-2093.1997. PMID 9169736
- [Background] Murdoch DA, Banatvaia N, Bone A, Shoismatulloev BI, Ward LR, Threlfall EJ. Epidemic ciprofloxacin-resistant Salmonella typhi in Tajikistan. Lancet. 1998 Jan 31;351(9099):339. doi: 10.1016/s0140-6736(05)78338-0. No abstract available. PMID 9652619
- [Derived] Szu SC, Lin KF, Hunt S, Chu C, Thinh ND. Phase I clinical trial of O-acetylated pectin conjugate, a plant polysaccharide based typhoid vaccine. Vaccine. 2014 May 7;32(22):2618-22. doi: 10.1016/j.vaccine.2014.03.023. Epub 2014 Mar 21. PMID 24657719